CLINICAL TRIAL: NCT04623190
Title: Using Health Information Technology to Improve Health Behaviors and Promote Cardiovascular Health Among Adolescent and Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202011075
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Disease; Young Adult Cancer Survivors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Providers (Experimental): -All eligible providers will be sent questionnaires electronically to their email at baseline and follow-up. Providers will be invited to attend a training session to educate them on the PREVENT tool at baseline. The providers will be delivering the PREVENT tool.
  Interventions: Behavioral: PREVENT tool
- Patients - Wait-List Control (Active Comparator): * Complete questionnaires and accelerometry at baseline (administered electronically or by mail; accelerometers administered by mail). Following baseline measurement, patients will be randomized and attend their clinic visit. Follow-up measures will be administered 3-months and 6-months after the clinic visit electronically and by mail
  * A PREVENT action plan (behavior change prescription, community resources, and education) will be provided to the patient via email after the completion of the follow-up measurement.
  Interventions: Behavioral: Wait-List Control
- Patients - PREVENT Tool (Experimental): * Complete questionnaires and accelerometry at baseline (administered electronically or by mail; accelerometers administered by mail). Following baseline measurement, patients will be randomized and attend their clinic visit. Follow-up measures will be administered 3-months and 6-months after the clinic visit electronically and by mail
  * At the clinic visit, the provider will use PREVENT tool to discuss risk and deliver a tailored behavioral change plan inclusive of patient-centered community resources. PREVENT will calculate patient's overall risk for developing cardiovascular disease. Physical activity and food intake recommendations are tailored to current weight status and health behaviors using evidence-based recommendations.
  Interventions: Behavioral: PREVENT tool

INTERVENTIONS:
Behavioral: Wait-List Control — -Will receive routine clinical care. After completion of follow-up measures, control participants will receive a behavior change prescription via the PREVENT tool
  Arms: Patients - Wait-List Control
Behavioral: PREVENT tool — -PREVENT is a novel Health Information Technology tool designed to promote physical activity and healthy food intake among overweight/obese patients at the point of care. PREVENT automates the delivery of personalized, evidence-based behavior change recommendations and provides an interactive map of community resources to help providers link patients to resources in their community.
  Arms: Patients - PREVENT Tool; Providers

SUMMARY:
Health information technology (HIT) has the potential to improve the quality, efficiency, consistency, and availability of cancer survivor care. PREVENT is a novel HIT tool designed by our team for adolescents (12-19 years). PREVENT aggregates and displays the American Heart Association's (AHA) Life Simple 7 cardiovascular health (CVH) risk factors and provides tailored, evidence-based, behavior change recommendations inclusive of community resources that are delivered to overweight/obese adolescents at the point-of-care to improve CVH. The investigators seek to expand this tool for patients beyond 19 years of age to increase this tool's reach to the entire adolescent and young adult (AYA) age range and then evaluate its effectiveness among AYA cancer survivors.

ELIGIBILITY:
Patient eligibility criteria

* Aged 20-39 years
* Prior diagnosis of pediatric cancer (diagnosed <21 years of age).
* Not receiving active therapy for their cancer
* Receiving care from the Pediatric Hematology/Oncology staff and physicians at St. Louis Children's Hospital, the St. Louis Children's Specialty Care Center, Siteman Cancer Center's Lifelong Outcomes Clinic at Siteman South County
* At risk for poor CVH (BMI ≥ 25 kg/m^2)
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Provider eligibility criteria.

-All providers and clinic staff (physicians, nurses, clinic staff, clinic research associates) in the Pediatric Hematology/Oncology program at St. Louis Children's Hospital and the CSCC or in the Siteman Cancer Center's Lifelong Outcomes Clinic at Siteman South County are eligible to participate.

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Change in minutes of physical activity | At baseline and 3-months
  Physical activity will be measured using a triaxial accelerometer (Actigraph GT3X+, Actigraph of Ft. Walton Beach, FL). The participant will be instructed to wear the accelerometer on an elasticized belt, on the left mid-axillary line. The Actigraph is one of the most common accelerometers used for scientific purposes. Participants will be encouraged to wear the accelerometer 24-hours per day for at least 7-days, including 2 weekend days.
Change in food intake behaviors | At baseline and 3-months
  Patient-reported food intake behaviors (fruit and vegetable intake, whole grains, sugar-sweetened beverages and snacking behaviors) are collected using a brief Health Behavior & Attitudes Survey.
Change in body mass index (BMI) | At baseline and 3-months
  Collected from patient's medical record.
Change on patient's attitudes toward behavior change | At baseline and 3-months
  A survey (6-question) administered to patients will assess attitudes toward and readiness for behavior change. Questions are asked using a 5-point Likert scale (range: 0-30) with a higher score indicating more positive attitudes.

SECONDARY OUTCOMES:
Change in patients' satisfaction of PREVENT tool: survey | Within 48 hours of clinic visit and at 3-months
Provider's satisfaction of PREVENT tool: survey | 3-months
  A survey (15-questions) will assess provider's satisfaction with five aspects of health information technology: content, accuracy, format, ease of use and timeliness. Questions are asked on a 5-point Likert scale (range: 15-75) with a higher score indicating greater satisfaction
Change on patient's average systolic and diastolic blood pressure | At baseline and 3-months
  Collected from patient's medical record
Change in patient's cholesterol | At baseline and 3-months
  Collected from patient's medical record
Change in patient's fasting blood glucose | At baseline and 3-months
  Collected from patient's medical record
Provider's motivation for sustained use of PREVENT tool | 3-months
  -A survey (12-questions) will assess provider's intent to change their behavior and continue using PREVENT were adapted from Legare's CPD Reaction Questionnaire. Questions are asked using a 7-point Likert scale (range: 12-84) with a higher score indicating greater motivation for sustained use.
Fidelity of PREVENT tool implementation | 0-3 months
  -Fidelity will be measured using direct observation of patient-provider interactions while using the PREVENT tool. A direct observation checklist will be used by the observer to determine the number of interactions with the PREVENT tool that were implemented as intended.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Kepper, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu